CLINICAL TRIAL: NCT02370420
Title: Intra-Articular Injections of Platelet-Rich Plasma in Knee Osteoarthritis: Unique Application Versus Triple Application
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Universidad Autonoma de Nuevo Leon (Other)
Responsible Party: Principal Investigator, FELIX VILCHEZ CAVAZOS, Dr. med. Jose Felix Vilchez Cavazos, Universidad Autonoma de Nuevo Leon
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OR15-002
Record Dates: First submitted 2015-01-27; First posted 2015-02-25 (Estimated); Results first posted 2018-02-19 (Actual); Last update posted 2018-02-19 (Actual); Status verified 2017-08

CONDITIONS: Osteoarthritis
Keywords: Platelet-rich plasma; Osteoarthritis
MeSH Terms: conditions — Osteoarthritis | interventions — Exercise Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Unique application of PRP (Experimental): Patients will be applied a unique application of platelet-rich plasma for knee osteoarthritis, and will be given rehabilitation exercises at home
  Interventions: Biological: Platelet-Rich Plasma; Behavioral: rehabilitation exercises
- Triple application of PRP (Active Comparator): Patients will be applied a triple application of platelet-rich plasma for knee osteoarthritis, with a interval of two weeks between each, and will be given rehabilitation exercises at home
  Interventions: Biological: Platelet-Rich Plasma; Behavioral: rehabilitation exercises

INTERVENTIONS:
Biological: Platelet-Rich Plasma — Autologous Platelet-Rich Plasma will be applied by a intra-articular injections
Behavioral: rehabilitation exercises — Patients would been shown rehabilitation exercises, to perform them at home

SUMMARY:
The investigators include patients attending the outpatient clinic in the area of Orthopedics and Traumatology of the investigators hospital with a diagnosis of knee osteoarthritis, which treatment is medical. Patients will be divided into two groups. In both groups, they will be given verbal, clear and detailed information on the approach to follow, the intra-articular application of Platelet-Rich Plasma in the knee, plus rehabilitation exercises. In the first group will be held single application, while in the second group three applications will be made at an interval of two weeks each. Both groups will be assessed before and after application, together with outpatient follow-up by the SF-12 Health Survey (SF-12), Western Ontario and McMaster Universities Arthritis Index (WOMAC) and Visual Analogue Scale (VAS).

DETAILED DESCRIPTION:
Osteoarthritis (OA ) refers to a clinical syndrome of joint pain with a multifactorial etiology , with the gradual loss of articular cartilage, osteophytosis formation, subchondral bone remodeling and inflammation of the joint. Is the most common cause of knee pain, and one of the leading causes of disability and dependence of the adult population that generates large expenditures in the area of health.

The clinical diagnosis of OA is primarily clinical - radiological, based on a complete medical history and physical examination directed. No laboratory studies are routinely requested since there is no specific diagnostic test or pathognomonic for diagnosis. Physical examination is most important.

The ideal treatment is a multidisciplinary one, and must meet the objectives of achieving anesthesia, reduce disability and improve joint function and patient's quality life, with low toxicity of drugs. Several conservative treatments are recommended by clinical guidelines. Some nonpharmacologic measures are: patient education, exercise, weight loss, modification of footwear, using the local cryotherapy, acupuncture and electromagnetic therapy. Drug therapy can be summarized in paracetamol, NSAIDs, opioids, and slow-acting drugs. If these oral drugs do not work can be administered intra-articularly (corticosteroids, viscosupplementation products, and blood derivates).

Platelet-Rich Plasma (PRP) is a rich source of growth factors such as Platelet-derived growth factor (PDGF), transforming growth factor β (TGF- β ), vascular endothelial growth factor (VEGF), like growth factor type I insulin (IGF- I), vascular endothelial growth factor (EGF), among others. For these growth factors are released, the platelets need to be activated by substances such as calcium chloride, calcium gluconate or thrombin. Once activated , growth factors are secreted, reaching a peak concentration 10 minutes. It is known that GF, PDGF and TGF -B stimulate chondrogenesis helping solving clinical manifestations of patients studied.

The investigators include patients attending the outpatient clinic in the area of Orthopedics and Traumatology of our hospital with a diagnosis of knee osteoarthritis, which treatment is medical. Patients will be divided into two groups. In both groups, they will be given verbal, clear and detailed information on the approach to follow, the intra-articular application of Platelet-Rich Plasma in the knee, plus rehabilitation exercises. In the first group will be held single application, while in the second group three applications will be made at an interval of two weeks each. Both groups will be assessed before and after application, together with outpatient follow-up by the SF-12, WOMAC and Visual Analogue Scale.

The PRP would be obtained through previous an asepsis and antisepsis of the patient's arm, 30cc of blood form the Basilic vein would be extracted.

Each sample will initially centrifuged at 1800 rpm for 10 minutes in a centrifuge and the sample would be separated into three layers : 1- Red Cell (lower) White 2- (plasma rich in growth factors) Yellow 3- ( plasma poor in growth factors ).1000 ul PRP ( yellow layer ) is extracted by placing it in 15 mL Falcon tubes for subsequently performing a second step of centrifugation at 3400 rpm for 12 minutes. The top layer of platelet poor plasma is removed and stayed with the lower layer, the PRP (3-5 mL ) . Before application in the patient's knee,calcium gluconate 10% was added, 0.15 mL per milliliter of PRP obtained. The sample then would be aspirated with a 10 mL syringe for the application to the patient.

After asepsis and antisepsis of where the puncture site , sterile drapes were placed clearing the workspace, the PRP is injected with a technique 45 ° at the corner superior- lateral patellar, reaching the joint capsule. Once injected the PRP, a sterile pad on the application area will be placed.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 90 years
* Patients with no previous treatment
* Patients with Knee osteoarthritis grade 1-2 ( Kellgren-Lawrence based on radiographic findings)

Exclusion Criteria:

* Age <18 and > 90 years
* Patients with Knee osteoarthritis grade 3-4 ( Kellgren-Lawrence based on radiographic findings)
* Patients with asociated Rheumatic syndromes
* Patients with anticoagulant therapy
* Patients with hepatic problems, Diabetes Mellitus, Coagulopathy, hearth conditions, immunodepressed, or infections
* Pregnant patients
* Patients with prosthetic or orthotic.
* Patients with hemoglobin values < 11g/dl , platelets < 150,000/μL

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Felix Vilchez, MD, PHD, Principal Investigator — Universidad Autonoma de Nuevo Leon
Locations (1):
- Facultad de Medicina UANL, Monterrey, Nuevo León, Mexico

REFERENCES:
- [Result] Martel-Pelletier J, Boileau C, Pelletier JP, Roughley PJ. Cartilage in normal and osteoarthritis conditions. Best Pract Res Clin Rheumatol. 2008 Apr;22(2):351-84. doi: 10.1016/j.berh.2008.02.001. PMID 18455690
- [Result] Jevsevar DS, Brown GA, Jones DL, Matzkin EG, Manner PA, Mooar P, Schousboe JT, Stovitz S, Sanders JO, Bozic KJ, Goldberg MJ, Martin WR 3rd, Cummins DS, Donnelly P, Woznica A, Gross L; American Academy of Orthopaedic Surgeons. The American Academy of Orthopaedic Surgeons evidence-based guideline on: treatment of osteoarthritis of the knee, 2nd edition. J Bone Joint Surg Am. 2013 Oct 16;95(20):1885-6. doi: 10.2106/00004623-201310160-00010. No abstract available. PMID 24288804
- [Result] Wang-Saegusa A, Cugat R, Ares O, Seijas R, Cusco X, Garcia-Balletbo M. Infiltration of plasma rich in growth factors for osteoarthritis of the knee short-term effects on function and quality of life. Arch Orthop Trauma Surg. 2011 Mar;131(3):311-7. doi: 10.1007/s00402-010-1167-3. Epub 2010 Aug 17. PMID 20714903
- [Result] Woolf AD, Pfleger B. Burden of major musculoskeletal conditions. Bull World Health Organ. 2003;81(9):646-56. Epub 2003 Nov 14. PMID 14710506
- [Result] Park SI, Lee HR, Kim S, Ahn MW, Do SH. Time-sequential modulation in expression of growth factors from platelet-rich plasma (PRP) on the chondrocyte cultures. Mol Cell Biochem. 2012 Feb;361(1-2):9-17. doi: 10.1007/s11010-011-1081-1. Epub 2011 Sep 29. PMID 21956670
- [Result] Kon E, Buda R, Filardo G, Di Martino A, Timoncini A, Cenacchi A, Fornasari PM, Giannini S, Marcacci M. Platelet-rich plasma: intra-articular knee injections produced favorable results on degenerative cartilage lesions. Knee Surg Sports Traumatol Arthrosc. 2010 Apr;18(4):472-9. doi: 10.1007/s00167-009-0940-8. Epub 2009 Oct 17. PMID 19838676

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The location of recruitment was the Orthopaedic and Traumatology consultation.
Pre-assignment Details: After the sign of the informed consent, the patients enrollment were assigned in the group of single injection or triple injection according to a randomization plan.
Period: Overall Study
Arm/Group | Unique Application of PRP | Triple Application of PRP
Started | 29 | 27
Completed | 15 | 15
Not Completed | 14 | 12
Not completed — Physician Decision | 3 | 3
Not completed — Lost to Follow-up | 11 | 9

BASELINE CHARACTERISTICS:
Population: The values were obtained only from the patients who completed the study and that were included in the final analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Unique Application of PRP | Triple Application of PRP | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 10 | 23
  >=65 years | 2 | 5 | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.46 (10.68) | 58.77 (11.19) | 56.61 (10.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 11 | 25
  Male | 1 | 4 | 5
Region of Enrollment [Number; unit: participants]
  Mexico | 15 | 15 | 30
Physical Component of the Short Form-12 of the Health Survey (SF-12) [Mean (Standard Deviation); unit: units on a scale] — We used the Spanish (México) version of the Short Form-12 of the Health Survey (SF-12) to assess the quality of life of the patient. This survey evaluates 2 main components: one physical and one mental, and each one is composed by 4 elements. The total value displayed represents the summatory of all the elements evaluated by the survey in the physical component.
  A higher value indicates a better quality of life. The scores range from 0 to 100. The data obtained with the SF-12 has been developed, tested and validated by Quality Metric Incorporated. Population: The values were obtained only form the patients who completed the study and that were included in the final analysis.
  units on a scale | 33.61 (9.14) | 37.25 (7.19) | 35.43 (8.18)
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) [Mean (Standard Deviation); unit: units on a scale] — We used the Western Ontario and McMaster Universities (WOMAC) Osteoarthritis Index to assess the overall clinical effectiveness of the two treatments. This index is composed by three categories: pain, articular stiffness, and functional limitation. The survey consists of 24 elements ranged from 0 (zero) to 4, with a higher value indicating a worst outcome. Thus, a reported value can range from 0 to 96. The values displayed correspond to the total WOMAC values integrated by the summatory of the three categories.
  units on a scale | 41.27 (19) | 41 (16.50) | 41.13 (17.75)
Visual Analog Scale (VAS) [Mean (Standard Deviation); unit: cm] — We used the Visual Analog Scale (VAS) to measure global pain on all patients. The scale used consisted on a 10 cm line divided in 10 equal parts. According to this, the possible values ranged from 0 (zero) to 10. The highest score (10) represented the highest level of pain.
  cm | 7.06 (2.21) | 6.46 (2.47) | 7.03 (2.34)

OUTCOME MEASURES:

1. Primary Outcome: Change in the Western Ontario and McMaster Universities (WOMAC) Ostearthritis Index (Therapeutic Effect)
Description: The Western Ontario and McMaster Universities (WOMAC) Osteoarthritis Index is a widely used, proprietary set of standardized questionnaires used by health professionals to evaluate the condition of patients with osteoarthritis of the knee and hip, including pain, stiffness, and physical functioning of the joints. It measures five items of pain (score range 0-20), two for stiffness (score range 0-8), and 17 for functional limitation (score range 0-68); thus, the total score range is 0-96. A higher value indicates a worst outcome.
  Only the final measures (at 24 weeks) are presented as part of the final analysis.
Time Frame: Baseline,3 weeks, 6 weeks, 12 weeks, 24 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Unique Application of PRP | Triple Application of PRP
Number analyzed (Participants) | 15 | 15
units on a scale | 28.53 (14) | 22.27 (19.07)

2. Secondary Outcome: Change in the SF-12 Health Survey (Quality of Life)
Description: SF-12 scale is a generic, multipurpose short-form survey with 12 questions selected from the SF-36 Health Survey which, when combined, scored and weighted, results in two scales of mental and physical functioning and overall health-related quality of life.
  A higher value indicates a better quality of life of the patient. The scores range from 0 to 100. The data obtained with the SF-12 has been developed, tested and validated by Quality Metric Incorporated.
  Only the final measures (at 24 weeks) from the physical domain are presented as part of the final analysis.
Time Frame: Baseline,3 weeks, 6 weeks, 12 weeks, 24 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Unique Application of PRP | Triple Application of PRP
Number analyzed (Participants) | 15 | 15
units on a scale | 41.79 (6.71) | 44.74 (10.65)

3. Secondary Outcome: Change in the Visual Analog Scale (VAS) (Global Pain)
Description: The Visual Analog Scale (VAS) is a unidimensional measure of pain intensity. The scale is most commonly anchored by "no pain " (score of 0) and "pain as bad as it could be" or "worst imaginable pain" (score of 10).
  Only the final measures (at 24 weeks) are presented as part of the final analysis.
Time Frame: Baseline,3 weeks, 6 weeks, 12 weeks, 24 weeks
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Unique Application of PRP | Triple Application of PRP
Number analyzed (Participants) | 15 | 15
cm | 4.46 (2.06) | 3.26 (3.12)

ADVERSE EVENTS:
Time Frame: Six months
Description: All patients were asked and evaluated for possibles adverse events at time-points of evaluation (most commonly pain at the site of injection). Specific attention was provided for platelet-rich plasma (PRP) treated patients.
Arm/Group | Triple Application of PRP | Unique Application of PRP
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 1/15 | 1/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Triple Application of PRP (N=15) | Unique Application of PRP (N=15)
Pain, inflammation (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) — Patients showing pain and inflammation at the site of the injection after they were treated with PRP. These symptoms prevailed for 48 hours after injection with spontaneous resolution.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No